CLINICAL TRIAL: NCT00006495
Title: Augmentation of HIV-Specific Helper and CTL Responses Through Therapeutic Vaccination in Individuals Receiving Potent Suppressive Antiretroviral Therapies
Brief Title: Immune Responses in HIV-Positive Patients Receiving an Anti-HIV Drug Combination When Given the HIV Vaccines Remune and vCP1452
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: Double | Purpose: Treatment
Other Study IDs: A5058s; 10674 (Registry Identifier: DAIDS ES Registry Number); ACTG A5058s; AACTG A5058s
Record Dates: First submitted 2000-11-15; First posted 2001-08-31 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Placebos; T-Lymphocytes, Helper-Inducer; AIDS Vaccines; RNA, Viral; HIV Core Protein p24; T-Lymphocytes, Cytotoxic; Anti-HIV Agents; HIV Therapeutic Vaccine
MeSH Terms: conditions — HIV Infections | interventions — HIV-1 immunogen, incomplete Freund's adjuvant

INTERVENTIONS:
Biological: ALVAC(2)120(B,MN)GNP (vCP1452)
Biological: HIV-1 Immunogen

SUMMARY:
The purpose of this study is to see how the vaccines Remune (HIV-1 immunogen) and vCP1452 affect immune responses in patients who also are taking anti-HIV medications. This study also will see if these vaccines are safe to use either alone or in combination.

Treatment with anti-HIV drugs does not always keep HIV viral load low and under control. This study will look at the effect of the HIV vaccine, vCP1452, on the immune response and how it works in combination with Remune. Information about immune responses and the safety of these vaccines in HIV-positive patients will be gathered.

DETAILED DESCRIPTION:
Human viral infections are controlled by the immune system. However, the multiple immune responses provoked by HIV infection do not control the infection in most people. The ability to specifically augment CTL responses with an immunotherapeutic vaccine may strengthen the containment of viremia afforded by antiretroviral agents and thereby extend the durability of viral suppression. The current study will attempt to determine whether therapeutic immunizations with HIV-1 immunogen and vCP1452 are safe and able to augment HIV-1 specific immune responses for a longer period of time than antiretroviral therapy alone, and if both agents are better than either by itself.

Patients currently enrolled in A5058s under A5057/A5058s Versions 1.0 and 2.0 will be given the option of continuing their participation in A5058s through this independent study. Rollover patients register to Step II and begin treatment/evaluations on A5058s at the same study week that they were on in Versions 1.0 and 2.0 of A5057/A5058s. New patients enter Step I and will not need to register to Step II. Step I patients are stratified on the basis of HIV viral load, antiretroviral history, and current antiretroviral treatment. Within each stratum, patients are randomized to 1 of the following 4 treatment arms: HIV-1 immunogen plus ALVAC placebo, HIV-1 immunogen placebo plus ALVAC placebo, HIV-1 immunogen placebo plus vCP1452, or HIV-1 immunogen plus vCP1452. Patients receive an injection at study entry and every 12 weeks thereafter until the end of the study, a minimum of 2 years. Step II patients receive the same treatment as patients in Step I. Patients are evaluated every 12 weeks for clinical, immunologic, and virologic parameters. Patients continue taking the antiretroviral treatment that they were taking at study entry until reaching a virologic relapse as defined in the protocol. If no response to a new drug regimen occurs, or the antiretroviral therapy is not changed, immunizations may continue as long as the viral load remains below 5,000 copies/ml.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for Step I of this study if they:

* Are at least 18 years old.
* Are HIV-infected.
* Have been on stable anti-HIV combination drug therapy for at least 12 weeks prior to screening for viral load and are willing to continue the same treatment during the study unless they experience side effects from the drugs and have a viral load increase.
* Have a viral load lower than 50 copies/ml at screening. Patients must have had a viral load below 500 copies/ml for at least 12 weeks prior to screening.
* Have a CD4 T cell count of at least 300 cells/mm3 within 30 days prior to study entry.
* Agree to practice acceptable methods of birth control, including male and female condoms, a diaphragm, or an intra-uterine device (IUD), while on study treatment and for 12 weeks after study treatment is discontinued.
* Patients may be eligible for Step II of this study if they:
* Are enrolled in A5058s under A5057/A5058s, Versions 1.0 and 2.0.

Exclusion Criteria

Patients will not be eligible for Step I of this study if they:

* Are pregnant or breast-feeding.
* Have an acute infection requiring antibiotics, an outbreak of a herpes virus, or other illness or surgery within 30 days prior to entry.
* Have a long-term infection other than HIV.
* Have cancer that may require systemic treatment.
* Have had lymph node irradiation.
* Have received any HIV vaccine.
* Have used GM-CSF, G-CSF, M-CSF, IFN, IL-2, or similar medication within 30 days prior to entry.
* Have used drugs affecting the immune system within 30 days prior to entry, or have an illness that may require use of these drugs.
* Have had immunizations within 30 days prior to study entry.
* Have received hydroxyurea within 30 days prior to study entry.
* Are allergic to egg proteins or neomycin or have had other serious allergic reactions.
* Work in close contact with canaries, or react to canarypox. Persons with a pet canary are not excluded.
* Have had 2 viral load measurements in a row taken at least 14 days apart that were 500 copies/ml or higher in the 12 weeks prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Study Completion 2004-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Spyros Kalams, Study Chair; Fred Valentine, Study Chair
Locations (9):
- United States (9):
  - UCLA CARE Center CRS, Los Angeles, California
  - Univ. of Miami AIDS CRS, Miami, Florida
  - Johns Hopkins Adult AIDS CRS, Baltimore, Maryland
  - Massachusetts General Hospital ACTG CRS, Boston, Massachusetts
  - Beth Israel Deaconess Med. Ctr., ACTG CRS, Boston, Massachusetts
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - Unc Aids Crs, Chapel Hill, North Carolina
  - Hosp. of the Univ. of Pennsylvania CRS, Philadelphia, Pennsylvania
  - Univ. of Texas Medical Branch, ACTU, Galveston, Texas